CLINICAL TRIAL: NCT06282393
Title: The FibriCheck Data Registry
Brief Title: FibriCheck Data Registry
Acronym: FDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qompium NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Z-2023072
Record Dates: First submitted 2024-02-08; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cardiac Arrhythmia
Keywords: Photoplethysmography; Single-lead electrocardiography
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FibriCheck recordings (Other)
  Interventions: Device: FibriCheck recordings

INTERVENTIONS:
Device: FibriCheck recordings — PPG and single-lead ECG measurements

SUMMARY:
The goal of this interventional clinical trial is to establish a comprehensive, structured database that includes photoplethysmography (PPG) measurements with simultaneously recorded electrocardiography (ECG) data to evaluate the FibriCheck Algorithm in patients with heart rhythm disorders.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Access to a smartphone to perform daily measurements
* Ability to understand Dutch
* Atrial Fibrillation diagnosis OR one of the following:

  * CHA2DS2-VASc score ≥2 (male) or ≥3 (female)
  * Underwent elective cardiac surgery
  * Known with:

    * Chronic obstructive pulmonary disease
    * Obstructive sleep apnea
    * Heart Failure
    * Hypertension
    * Previous stroke or transient ischaemic attack
  * Having palpitations and/or racing heart as symptoms
  * Other arrhythmia such as atrial flutter, premature atrial contractions (PAC), premature ventricular contractions (PVC)

Exclusion Criteria:

* Individuals which are currently in follow-up with their physician, using the FibriCheck application
* Individuals with unnaturally coloured fingers (i.e. tattoos, ink); this may weaken the signal and may interfere with the effectiveness of the device
* Persons with conditions causing tremors or the inability to hold their hand still for at least 60 seconds (e.g. Parkinson or dementia) as, in this case, the device may not be able to accurately process a measurement
* Persons with reduced blood flow in the fingertips (e.g. perniosis or severe callus formation) as the device may not be able to detect the intensity variations induced by the blood flow
* Persons that have a disability to perform the measurements according to the instructions for use
* Persons with cardiac pacemakers, implantable cardioverter-defibrillators, or other implanted electronic devices as these can control the natural heart rhythm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Alignment PPG measurement | 14 days
  ECG-PPG alignment (RR-intervals)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Vandervoort, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium